CLINICAL TRIAL: NCT05620290
Title: MRI-Guided Focused Ultrasound Radiosensitization for Patients With Malignant Melanoma and Non Melanoma Skin Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Terry Fox Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4877
Record Dates: First submitted 2022-05-17; First posted 2022-11-17 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-12

CONDITIONS: Melanoma
Keywords: Focused ultrasound; Melanoma; Microbubbles
MeSH Terms: conditions — Melanoma | interventions — perflutren

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Arm (Experimental): Malignant Melanoma patients undergoing MRI-guided ultrasound-stimulated microbubble treatment plus radiation therapy
  Interventions: Drug: Definity; Device: Sonalleve Focused Ultrasound Device

INTERVENTIONS:
Drug: Definity — Stimulation of Definity microbubbles using Sonalleve device within tumour vasculature
Device: Sonalleve Focused Ultrasound Device — Sonalleve Focused Ultrasound Device

SUMMARY:
The objective of this study is to examine the safety profile and therapeutic efficacy of MRI-guided focused ultrasound microbubble therapy and radiotherapy in humans.

DETAILED DESCRIPTION:
The approach uses relatively low-power ultrasound, operating with lower power levels than high intensity focused ultrasound and ultrasound-based hyperthermia techniques, delivered on the Sonalleve platform. The tumour will be sonicated before the radiation to enhance the effect of therapy. The technique is spatially targeted and stimulates microbubbles using low-power ultrasonic fields in the tumour location only. the primary aim of this research is to evaluate the safety profile of MRI-guided ultrasound stimulated microbubble treatment and radiation in patients with malignant melanoma. The secondary aim is to evaluate tumour (primary and/or metastasis) response to MRI-guided ultrasound stimulated microbubble treatment and radiation, as measured radiologically within the treated regions.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* All biopsy-confirmed malignant melanoma of the skin and non melanoma skin cancer, including metastatic lesions.
* Stage I-IV malignant melanoma and non melanoma skin cancer, per AJCC guidelines (8th Edition).
* Patient referred for palliative radiotherapy/ standard radiotherapy/ neoadjuvant radiotherapy/ SBRT/ hypofractionation.
* Patient on immunotherapy.
* Able to understand and give informed consent. Weight <140kg.
* Target lesion visible by non-contrast MRI.
* Target lesion accessible for MRg-FU procedure.
* Able to communicate sensation during MRg-FU treatment.
* Creatinine within normal institutional limits or creatinine clearance >60 mL/min/1.73 m2 for patients with creatinine levels above the institutional upper limit of norma

Exclusion Criteria:

* Pregnant or lactating women may not participate due to the embryotoxic effects of protocol treatment. Women/ men of reproductive potential may not participate unless they have agreed to use an effective contraceptive method.
* Unable to have contrast-enhanced MRI scan - the standard of care criteria
* Target lesion involves the skin surface causing ulceration, bleeding or discharge
* Severe cardiovascular, neurological, renal or hematological chronic disease
* ECOG (Eastern Cooperative Oncology Group) Performance Status ≥ 3. Unable to tolerate required stationary position during treatment
* Cardiac disease or unstable hemodynamics, including myocardial infarction within six months, unstable angina, congestive heart failure, ejection fraction < 50%, cardiac shunts, cardiac arrhythmia and cardiac pacemaker.
* Contraindication to perflutren including subjects with a family or personal history of QT prolongation or taking concomitant medications known to cause QTc prolongation like cisapride, erythromycin, tricyclic antidepressants, Class IA and III antiarrhythmic agents and some antipsychotics like haloperidol, droperidol, quetiapine, thioridazine, ziprasidone.
* Severe hypertension (diastolic BP > 100 mmHg)
* History of bleeding disorder, coagulopathy
* Severely impaired renal function with estimated glomerular filtration rate < 30ml/min/1.73m2 and/or on dialysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-06-15 (Actual); Primary Completion 2025-07-11 (Estimated); Study Completion 2028-07-11 (Estimated)

PRIMARY OUTCOMES:
Incidence of toxicity and adverse events, scored on the National Cancer Institute Common Toxicity Criteria (NCI CTCAE 4.03) | 90 days
  The patient will be assessed by a physician investigator and clinical research assistant (CRA) on the MRI-guided focused ultrasound + microbubble (MRgFUS + MB) treatment date and within follow up period of 90 days after treatment.

SECONDARY OUTCOMES:
Radiological response | 2 years
  The secondary aim is to evaluate tumour (primary and/or metastasis) response to MRgFUS + MB and radiation, which will be evaluated by tumour volume change.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Gregory Czarnota, MD, Ph.D., Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No